CLINICAL TRIAL: NCT05084079
Title: The Impact of Different Initial Insulin Dose Regimens on Time to Achieve Glycemic Targets and Treatment Safety in Short-term Intensive Insulin Therapy(SIIT)
Brief Title: Different Initial Insulin Dose Regimens on Time to Achieve Glycemic Targets and Treatment Safety in SIIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, Director of Endocrinology and Metabolism Department, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021526
Record Dates: First submitted 2021-09-26; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases
Keywords: Short-term intensive insulin therapy; Insulin dose; Time to glycemic goal; Hypoglycemic; Glycemic variability
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Formula-based (Experimental): Initial insulin regimen was decided according to the formula developed by the investigators previously.
  Interventions: Drug: CSII with formula-based initial insulin regimen
- Weight-based (Placebo Comparator): Initial insulin regimen was decided according to current guidelines.
  Interventions: Drug: CSII with weight-based initial insulin regimen

INTERVENTIONS:
Drug: CSII with formula-based initial insulin regimen — Initial total daily insulin dose(TDD) for CSII was calculated with a formula :（estimate TDD-1(eTDD-1) = 0.35× body weight (kg) + 2.05× FPG (mmol/L) + 4.24×triglyceride(mmol/L) + 0.55× waist circumference (cm) - 49.1）, 42% of which was assigned as total basal dose and 58% as total premeal dose, with the pre-meal doses divided into 30:35:35 for breakfast, lunch and dinner.
  Other Names: Formula-based regimen
  Arms: Formula-based
Drug: CSII with weight-based initial insulin regimen — TDD for CSII was started with 0.5 IU/kg, 50% of which was assigned as total basal dose and 50% as total premeal dose, and the total pre-meal dose was divided equally before each meal.
  Other Names: Weight-based regimen
  Arms: Weight-based

SUMMARY:
To compare the effects of different initial insulin dose regimens during the short-term insulin intensive treatment on time to glycemic goal, hypoglycemia prevalence, glycemic variability and other safety problems in newly diagnosed type 2 diabetes mellitus(T2DM) patients, in order to investigate the rational of formula based initiation regimen.

DETAILED DESCRIPTION:
Diabetes has become one of the major chronic non-communicable diseases. Its prevalence was rising in these years. Short-term intensive insulin therapy can improve the β-cell function and nearly half of the patients can live with long-term glycemic remission. It has therefore become the recommended treatment for the newly diagnosis T2DM patients with high blood glucose. However, due to the glycemic goal for intensive therapy is strict, it's important to find out a suitable initial insulin regimen for continuous subcutaneous insulin infusion(CSII) with which patients can achieve euglycemia safely, stably and rapidly. In previous study, the investigators found out that the total daily insulin dose at the first day when euglycemia was achieved（TDD-1） was associated with weight, waist circumference, triglycerides and fasting blood glucose levels. According to this, the investigators figured out a formula for estimation of insulin dose for the short-term intensive insulin therapy in patients with newly diagnosed T2DM. However, its feasibility needs to be further verified. Therefore, the investigators conducted this prospective randomized controlled study to compare the effects of different initial insulin dose regimens during the short-term insulin intensive treatment on time to glycemic goal, hypoglycemia prevalence, glycemic variability and other safety problems in newly diagnosed type 2 diabetes patients, in order to investigate the rational of formula based initiation regimen.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes (1999 World Health Organization standard);
* Type 2 diabetic patients who have never received any hypoglycemic therapy (including oral hypoglycemic agents, Chinese medicine , and insulin);
* Body mass index (BMI) between 20-35 kg/m2;
* Fasting plasma glucose (FPG) levels between 7.0 -16.7 mmol/L, glycated haemoglobin >7.0%;
* Willing to receive CSII intensive treatment during hospitalization and monitoring blood glucose 8 times per day.

Exclusion Criteria:

* Type 1 diabetes or special type of diabetes;
* Acute complications of diabetes: ketoacidosis, hyperosmolar coma, lactic acidosis, etc.;
* Severe macrovascular complications: acute cerebral vascular accidents, acute coronary syndromes, peripheral arterial disease requiring vascular intervention or amputees for hospitalization occur within 12 months before selection;
* Severe microvascular complications: proliferative phase retinopathy; urinary albumin excretion rate(AER)> 300 mg/g or urinary protein Positive, quantitative> 0.5 g/d; uncontrolled painful diabetic neuropathy and significant diabetic autonomic neuropathy;
* Obvious liver and kidney dysfunction: alanine aminotransferase ≥ 2.5 times the upper limit of normal, total bilirubin ≥ 1.5 times the upper limit of normal, serum creatinine greater than 150 umol/L or creatinine clearance less than 50 mL/min;
* Significant increase in blood pressure: blood pressure continued to be higher than 180/110 mmHg;
* Significant anemia: hemoglobin <100g /L may require regular blood transfusions;
* Use of drugs that may affect blood glucose during 12 weeks, such as oral/intravenous corticosteroids, growth hormone, estrogen/progestogen, high-dose diuretics, antipsychotics, etc. Low-dose diuretics for antihypertensive purposes (hydrochlorothiazide <25 mg/d, indapamide ≤ 1.5 mg/d), and physiological quantities of thyroid hormones used for replacement therapy are not limited to this;
* Effects associated with other underlying diseases influenced the observation of blood glucose, such as systemic infection or severe comorbidity, malignancy or chronic diarrhea, uncontrolled endocrine gland function abnormalities, chronic cardiac insufficiency (grade III and above), psychosis, or pregnant;
* The patients does not cooperate, or the investigator judges that it may be difficult to complete the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
The time to glycemic goal | 1 year
  After CSII begin, the time(days) to reach glycemic goal of each patients. The glycemic goal defined as at least six out of eight-point fingertip blood glucose meet the standard that fasting blood glucose(FBG) or non-postprandial blood glucose is between 4.4-6.0 mmol/L and 2h postprandial blood glucose(PBG) is between 4.4-8.0 mmol/L.

SECONDARY OUTCOMES:
Incidence of hypoglycemia | 1 year
  Differences in incidence of hypoglycemia among treatment arms at the end of study.
Change of blood glucose fluctuations | 1 year
  Differences in blood glucose fluctuations among treatment arms at the end of study.
Change of β cell function | 1 year
  Differences in β-cell indicators among treatment arms at the end of study.
Change of insulin sensitivity | 1 year
  Differences in insulin sensitivity indicators among treatment arms at the end of study.
Change of insulin dosage | 1 year
  Differences in insulin dosage among treatment arms at the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Li, MD,PhD, Principal Investigator — endocrinology department of the first affiliated hospital of Sun Yat-sen University
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Liu L, Ke W, Wan X, Zhang P, Cao X, Deng W, Li Y. Insulin requirement profiles of short-term intensive insulin therapy in patients with newly diagnosed type 2 diabetes and its association with long-term glycemic remission. Diabetes Res Clin Pract. 2015 May;108(2):250-7. doi: 10.1016/j.diabres.2015.02.011. Epub 2015 Feb 21. PMID 25765670